CLINICAL TRIAL: NCT01842802
Title: Clinical Investigation of Non Invasive Fat Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: CYN12-NIF-ABDM02
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Subcutaneous Fat
MeSH Terms: interventions — Lasers, Semiconductor; Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diode Laser Treatment Before Abdominoplasty (Experimental): Patient will be treated with Diode Laser prior to abdominoplasty.
  Interventions: Device: Diode Laser
- YAG Laser Treatment Before Abdominoplasty (Experimental): Patients will be treated with YAG prior to abdominoplasty
  Interventions: Device: YAG laser

INTERVENTIONS:
Device: Diode Laser — Diode Laser for treatment of subcutaneous fat
  Arms: Diode Laser Treatment Before Abdominoplasty
Device: YAG laser — YAG laser for treatment of subcutaneous fat
  Arms: YAG Laser Treatment Before Abdominoplasty

SUMMARY:
The purpose of this study is to compare non invasive treatments using a YAG and Didode Laser to reduce the volume of fat.

ELIGIBILITY:
Inclusion Criteria:

* A healthy non-smoking male or female between 20-60 years of age
* Subjects presenting excess abdominal tissue (fat and skin), are candidates for an abdominoplasty procedure and are willing to allow the use of this device on their skin
* Subjects who will allow the excess skin removed as part of the abdominoplasty to be sent for laboratory analysis
* Understand and accept the obligation associated with the procedure
* Subjects with Fitzpatrick skin types I to III.
* Subjects who are willing to consent to participate in the study will be asked to undergo biopsies, ultrasound measurements, and blood testing as outlined for each group and defined in section 6.0.
* Subjects must agree to maintain the same diet and exercise regime throughout the study

Exclusion Criteria:

* Any previous liposuction/lipo-sculpture or any type of procedure in the abdominal area in the past 6 months
* A history of allergic reactions to medications or anesthesia required for the procedure
* A history of thrombophlebitis
* A history of acute infections
* A history of heart failure
* Received or is anticipated to receive antiplatelets, anticoagulants, thrombolytics, vitamin E or anti-inflammatories within 2 weeks pre treatment
* Intolerance to anesthesia or medications to be prescribed before or after the procedure.
* Any medical condition, that, in the investigator's opinion would interfere with the patient's participation in the study including EMLA cream or percocet
* Taking medications that are photosensitive
* A history of keloid formation
* A study subject must not be pregnant or have been pregnant in the last 3 months
* The physician has the right to make determination of eligibility as he/she deems clinically significant based on standard of care treatment

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Biopsy of Tissue Samples as a Measure of Effectiveness | 5 months post treatment
  Biopsy of treated area will be obtained up to 5 months post treatment and will be histologically assessed for changes in adipocytes and surrounding tissue to determine effectiveness of device.
Ultrasound Measurement to Evaluate Reduction of Fat | 5 months post treatment
  Ultrasound of the treatment area will be performed and evaluated in comparison to baseline results to determine reduction of the subcutaneous fat layer.

SECONDARY OUTCOMES:
Lipid level blood testing to evaluate changes post treatment | 5 months post treatment
  Blood testing will be performed to evaluate changes in lipid levels post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Aesthetic Pavilion, Staten Island, New York, United States